CLINICAL TRIAL: NCT07243860
Title: The Impact of Neuromuscular Rehabilitation on Knee Function and Brain Plasticity in Patients With Anterior Cruciate Ligament Rupture and Reconstruction
Brief Title: Neuromuscular Rehab for ACL Reconstruction: Knee Function & Brain Plasticity
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M20250812
Record Dates: First submitted 2025-09-09; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-10

CONDITIONS: Anterior Cruciate Ligament Injuries
Keywords: Anterior Cruciate Ligament Injuries; Neuromuscular Training; Knee Function; Neuroplasticity
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neuromuscular Training (Experimental)
  Interventions: Behavioral: Neuromuscular Training
- Conventional Rehabilitation (Active Comparator)
  Interventions: Behavioral: Conventional Rehabilitation

INTERVENTIONS:
Behavioral: Neuromuscular Training — This is a structured, supervised neuromuscular training program designed to enhance sensorimotor control, strength, and functional stability of the knee joint. The program is administered by certified physical therapists and consists of three phases:
  1. Preoperative Phase (6 weeks):
  2. Postoperative Phase (0-12 weeks):
  3. Postoperative Phase (12+ weeks):
  Core components include:Proprioception and Balance Training；Strength Training；Plyometrics and Dynamic Stability；Movement Pattern Re-training.
  Dosage:Frequency: 3 supervised sessions per week. Duration: Each session lasts approximately 60 minutes. Total Program Length: Preoperative phase (6 weeks) + postoperative phase (continued until specific functional criteria are met, approximately 12weeks post-op).
  Arms: Neuromuscular Training
Behavioral: Conventional Rehabilitation — This arm receives the standard of care rehabilitation protocol, which mirrors the experimental group in duration, frequency, and timing but differs fundamentally in the content and specificity of the exercises.
  Core components include (across both pre-operative and post-operative phases):
  Range of Motion (ROM) Exercises;Basic Strength Training;Standard Balance Training
  Dosage (Identical in timing to the experimental group):
  Pre-operative Phase: 6 weeks of training. Post-operative Phase: Continues until standard discharge criteria are met. Frequency: 3 supervised physical therapy sessions per week. Duration: Each session lasts approximately 60 minutes. Total Program Length: Continues until standard discharge criteria are met (typically 12 weeks post-op).
  Arms: Conventional Rehabilitation

SUMMARY:
This study focuses on patients with anterior cruciate ligament (ACL) rupture and reconstruction, aiming to systematically investigate the clinical efficacy and underlying mechanisms of neuromuscular training in restoring knee joint function.Beyond examining improvements in local knee biomechanics, the research delves into brain plasticity changes during rehabilitation to reveal the central regulatory mechanisms of neuromuscular control.The findings are expected to provide a solid theoretical and empirical foundation for optimizing post-ACL rehabilitation strategies, fostering interdisciplinary integration from peripheral interventions to neural central regulation.

DETAILED DESCRIPTION:
In the field of sports medicine, anterior cruciate ligament (ACL) injury is a common yet severe sports-related condition with significant consequences. Patients exhibit considerable variation in knee functional recovery following anterior cruciate ligament reconstruction (ACLR). Although neuromuscular training serves as an effective rehabilitation intervention, its mechanistic underpinnings remain incompletely elucidated, and the relationship between brain plasticity and functional recovery of the knee joint has not been sufficiently explored. Therefore, this study focuses on patients with ACL rupture and reconstruction, aiming to elucidate the specific mechanisms through which neuromuscular training contributes to the restoration of neuromuscular function in patients following ACL rupture and reconstruction, with particular emphasis on its effects on brain plasticity and neuromuscular control. It will systematically investigate the dynamic changes in brain functional plasticity and their underlying mechanisms throughout the rehabilitation process post-ACL injury and reconstruction. By uncovering the operational mechanisms of neuromuscular training in injury prevention and rehabilitation, this research will provide new empirical evidence to advance the theoretical framework of sports rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

1. Body Mass Index (BMI) ≥18.5 kg/m² and <35 kg/m²;
2. Diagnosed with first-time, unilateral, isolated anterior cruciate ligament (ACL) rupture ;
3. No or only mild concomitant injuries to the posterior cruciate ligament, medial collateral ligament, or lateral collateral ligament;
4. Voluntarily participated in the study and provided written informed consent .

Exclusion Criteria:

1. Patients with ACL rupture for more than 6 months;
2. Combined severe injuries (Grade II or higher) to the posterior cruciate ligament, medial collateral ligament, or lateral collateral ligament(Grading Note: Grade II indicates partial tear with ligament thickening, tortuosity, and fiber disruption; Grade III indicates complete rupture);OR combined severe meniscal tears ;
3. History of prior knee surgery (e.g., meniscal repair, ligament reconstruction, arthroplasty, arthroscopic debridement);
4. Presence of other knee pathologies: knee osteoarthritis, tumors, rheumatoid arthritis, tuberculosis, infectious or inflammatory diseases, fractures, dislocations, or other skeletal injuries;
5. Severe cardiac, pulmonary, cerebral, hepatic, or renal dysfunction; OR visual/cognitive impairments.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
isokinetic muscle strength | Pre-intervention and preoperative intervention, at 12 weeks and 12 months postoperatively
  The isokinetic muscle strength test selected angular velocities of 60°/s (slow) and 180°/s (medium). Observe the peak torque of the quadriceps femoris and hamstring muscles, the relative peak torque, the limb symmetry index, the ratio of peak torque between the hamstring and quadriceps muscles, and the total work.
sEMG | Pre-intervention and preoperative intervention, at 12 weeks and 12 months postoperatively
  The American-made Delsys wireless surface EMG system was used to measure EMG signals from the lower limb muscles during walking, running, and single-leg standing. A total of five muscles on the affected lower limb were recorded, including the rectus femoris (RF), vastus lateralis (VL), vastus medialis (VM), biceps femoris (BF), and semitendinosus (ST).The parameters collected and analyzed using the Delsys surface electromyography (sEMG) system include: raw EMG values during walking, running, and single-leg standing，root mean square (RMS) amplitude.
Three-Dimensional Gait Analysis using the Vicon System | Pre-intervention and preoperative intervention, at 12 weeks and 12 months postoperatively
  During the running process, the joint angles and torques of the hip joint, knee joint and ankle joint in the sagittal plane, coronal plane and horizontal plane, as well as the peak vertical ground reaction force, vertical instantaneous loading rate and rate of internal knee extension moment
Electroencephalography Assessment | Pre-intervention and preoperative intervention, at 12 weeks and 12 months postoperatively
  Electroencephalogram (EEG) analysis involves extracting raw EEG data during motor tasks and performing domain-specific feature analyses. This includes power spectral density and relative power as frequency-domain metrics, as well as functional and effective connectivity measures such as coherence and Granger causality.

SECONDARY OUTCOMES:
IKDC 2000 | Pre-intervention and preoperative intervention, at 12 weeks and 12 months postoperatively
  The International Knee Documentation Committee (IKDC) 2000 Subjective Knee Form is a standardized tool for evaluating knee function, pain, and activity levels in patients with ligament injuries, meniscal tears, or osteoarthritis. It consists of 18 items assessing symptoms, sports participation, and quality of life, with scores ranging from 0 to 100 (higher scores indicate better function)
Lysholm Knee Score | Pre-intervention and preoperative intervention, at 12 weeks and 12 months postoperatively
  The Lysholm Knee Score is an 8-item questionnaire designed to quantify knee function, particularly for ligament injuries, meniscal tears, and patellofemoral disorders. It evaluates pain, instability, locking, swelling, and mobility (e.g., stair climbing, squatting), with a total score of 0-100 (higher scores reflect better outcomes).

IPD SHARING:
Plan to Share IPD: Yes